CLINICAL TRIAL: NCT07387133
Title: Early Childhood Parental Technoference and Behavioral-Emotional Development: A Six-Month Prospective Study
Brief Title: Parental Technoference and Behavioral-Emotional Development in Early Childhood: A 6-Month Prospective Study
Acronym: TECH-SDQ
Status: Not yet recruiting | Type: Observational
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Timucin imdadoglu, MD, Specialist in Pediatrics (MD), Saglik Bilimleri Universitesi
Other Study IDs: TEKNOFERANS-SDQ-2026; EthicsNo-2026/19-Sancaktepe (Other: Sancaktepe Şehit Prof. Dr. İlhan Varank Training and Research Hospital Ethics Committee)
Record Dates: First submitted 2026-01-27; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Parental Technoference; Child Behavioral Problems; Emotional Development in Early Childhood
Keywords: parent-child interaction; screen time; preschool children; Strengths and Difficulties Questionnaire; digital media use

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Parent-Child Dyads (24-60 Months): This cohort includes parents and their children aged 24 to 60 months who attend a pediatric outpatient clinic at a tertiary training and research hospital. Participants are assessed at baseline using questionnaires evaluating parental technoference, parental and child screen time, and children's behavioral and emotional characteristics. A follow-up assessment is conducted six months later. This is an observational study, and no intervention is assigned.

SUMMARY:
This study aims to examine the relationship between parental technoference (parents' use of smartphones or other digital devices while spending time with their children) and behavioral and emotional development in early childhood.

The study will include parents of children aged 24 to 60 months who attend a pediatric outpatient clinic. At the beginning of the study, parents will complete an online questionnaire that includes questions about their own smartphone screen time, their child's screen exposure, and standardized questionnaires assessing parental technoference and children's behavioral and emotional characteristics.

Six months after the initial assessment, parents will be contacted again to complete a short follow-up questionnaire, including the behavioral and emotional assessment. The study does not involve any medical intervention or experimental treatment. All participation is voluntary, and responses will be collected anonymously.

The findings of this study are expected to contribute to a better understanding of how parental digital device use during daily interactions may be associated with children's emotional and behavioral development in early childhood.

DETAILED DESCRIPTION:
This is a single-center, prospective observational study conducted among parents of children aged 24 to 60 months attending a pediatric outpatient clinic at a tertiary training and research hospital.

Parental technoference is defined as interruptions in parent-child interactions due to parental use of smartphones or other digital devices. At baseline, participating parents will complete an online questionnaire that includes sociodemographic characteristics, self-reported average daily smartphone screen time over the previous seven days (recorded from the device's built-in screen time or digital wellbeing function), and information about the child's daily screen exposure.

Parental technoference will be assessed using a validated parental technoference scale, and children's behavioral and emotional characteristics will be evaluated using the parent-report version of the Strengths and Difficulties Questionnaire (SDQ) for preschool-aged children. Both instruments have established validity and reliability in the Turkish population.

At the end of the baseline assessment, parents will be provided with a brief informational message aimed at increasing awareness of digital distractions during parent-child interactions. No behavioral intervention will be enforced as part of the study.

Six months after the initial assessment, parents will be re-contacted via phone or email and invited to complete a follow-up questionnaire, including the SDQ and updated information on parental and child screen exposure. The primary outcome is the association between parental technoference levels and children's behavioral and emotional outcomes. Secondary outcomes include changes in SDQ scores over the six-month follow-up period.

All data will be collected anonymously and analyzed using appropriate statistical methods, including correlation analyses and multivariable regression models. This study involves no medical intervention and poses minimal risk to participants.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 24 to 60 months.
* Parent or primary caregiver able to read and understand Turkish.
* Parent uses a smartphone and can access device-based screen time information.
* Ability to complete an online questionnaire.
* Provision of written informed consent by the parent or legal guardian.
* Availability for a 6-month follow-up assessment.

Exclusion Criteria:

* Children with severe neurodevelopmental disorders (e.g., autism spectrum disorder, severe intellectual disability, neurometabolic diseases).
* Parents unable to reliably complete questionnaires due to cognitive, psychiatric, or language-related limitations.
* Parents who do not use a smartphone or cannot access screen time data.
* Refusal or inability to provide informed consent.
* Inability to be contacted for follow-up assessment.

Ages: 24 Months to 60 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The study population consists of parents and their children aged 24 to 60 months who attend a pediatric outpatient clinic at a tertiary training and research hospital.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Child Behavioral and Emotional Difficulties (SDQ Total Difficulties Score) | Baseline and 6 months
  Children's behavioral and emotional difficulties will be assessed using the parent-report version of the Strengths and Difficulties Questionnaire (SDQ). The primary outcome is the SDQ Total Difficulties Score measured at baseline and at 6-month follow-up.

SECONDARY OUTCOMES:
Parental Technoference Level | Baseline
  Parental technoference will be measured using a validated parental technoference scale assessing the frequency of digital device-related interruptions during parent-child interactions.
Changes in Children's Behavioral and Emotional Characteristics Over Time | Baseline to 6 months
  Changes in children's behavioral and emotional characteristics will be evaluated by comparing SDQ Total Difficulties and subscale scores between baseline and the 6-month follow-up assessment.
Child Screen Exposure | Baseline and 6 months
  Child screen exposure will be assessed based on parent-reported average daily screen time across different digital media devices.

CONTACTS AND LOCATIONS:
Locations (1):
- Sancaktepe Prof. Dr. Ilhan Varank Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared, as the study involves anonymized questionnaire-based data collected for observational research purposes only, and no data sharing plan has been approved by the ethics committee.

REFERENCES:
- [Result] Moemenbellah-Fard MD, Shahriari B, Azizi K, Fakoorziba MR, Mohammadi J, Amin M. Faunal distribution of fleas and their blood-feeding preferences using enzyme-linked immunosorbent assays from farm animals and human shelters in a new rural region of southern Iran. J Parasit Dis. 2016 Mar;40(1):169-75. doi: 10.1007/s12639-014-0471-1. Epub 2014 May 25. PMID 27065620
- [Result] Goodman R. The Strengths and Difficulties Questionnaire: a research note. J Child Psychol Psychiatry. 1997 Jul;38(5):581-6. doi: 10.1111/j.1469-7610.1997.tb01545.x. PMID 9255702